CLINICAL TRIAL: NCT00406926
Title: The Effect of Recombinant Human Growth Hormone Treatment on the Growth of Infants and Toddlers With Turner Syndrome
Brief Title: The Effect of Growth Hormone in Very Young Girls With Turner Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2878; B9R-US-GDFG
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome | interventions — Human Growth Hormone

INTERVENTIONS:
Drug: Somatropin

SUMMARY:
This study investigated the effect of growth hormone on the growth of infants and toddlers with Turner syndrome during 2 years of treatment with growth hormone. This was compared with the growth of infants and toddlers with Turner syndrome who did not receive any growth hormone treatment. The overall aim was to prevent the growth failure usually seen during this period. The study also looked at middle ear disease, hearing problems, and cognitive and behavioral development.

ELIGIBILITY:
Inclusion Criteria:

* Karyotype-proven Turner syndrome that included a documented abnormality of the short arm of an X chromosome.
* At least 9 months of age and not greater than 4 years of age.
* Normal values for age for hemoglobin, thyroid stimulating hormone (TSH) and urinalysis (office dipstick is adequate), performed prior to study entry.
* If there was a known history of hypothyroidism, then adequate thyroid hormone replacement must have been taken for at least 6 months prior to study entry.

Exclusion Criteria:

* Current or previous treatment with any therapy that may have directly influenced growth, including growth hormone, growth hormone-releasing hormone, estrogens and anabolic steroids such as oxandrolone. This included previous completion of, or withdrawal from, this study or any other study investigating therapeutic uses of growth hormone or growth hormone-releasing hormone.
* Chronic treatment with systemic glucocorticoids in supra-physiological doses.
* Treatment with potential growth-influencing medications such as methylphenidate (Ritalin), pemoline (Cylert), and amphetamines, at, or within 3 months prior to, study entry.
* Presence of any Y chromosome component in the karyotype if gonads were in situ. Subjects whose karyotype contained Y chromatin, but who had undergone gonadectomy, were eligible to enter the study.
* Presence of any additional known autosomal abnormality.

Ages: 9 Months to 4 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 1999-08; Study Completion 2003-08

PRIMARY OUTCOMES:
Height at the end of two years in the study.

SECONDARY OUTCOMES:
Middle ear problems assessed every 4 months
Hearing problems assessed annually
Cognitive and behavioral development assessed annually

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stanford, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hartford, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington